CLINICAL TRIAL: NCT05966272
Title: A Multi-center, Randomized, Double-blind, Placebo- Parallel Controlled, Phase II Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Type 2 Diabetes Subjects
Brief Title: Efficacy and Safety of HRS9531 Injection in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-202
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A multi-center, randomized, double-blind, placebo- parallel controlled Phase II clinical study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group A (Experimental): HRS9531 injection dose level 1
  Interventions: Drug: HRS9531 injection
- Treatment group B (Experimental): HRS9531 injection dose level 2
  Interventions: Drug: HRS9531 injection
- Treatment group C (Experimental): HRS9531 injection dose level 3
  Interventions: Drug: HRS9531 injection
- Treatment group D (Experimental): HRS9531 injection dose level 4
  Interventions: Drug: HRS9531 injection
- Treatment group E (Placebo Comparator): HRS9531 injection Placebo dose level 1
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group F (Placebo Comparator): HRS9531 injection Placebo dose level 2
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group G (Placebo Comparator): HRS9531 injection Placebo dose level 3
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group H (Placebo Comparator): HRS9531 injection Placebo dose level 4
  Interventions: Drug: HRS9531 injection Placebo

INTERVENTIONS:
Drug: HRS9531 injection — single dose
  Arms: Treatment group A; Treatment group B; Treatment group C; Treatment group D
Drug: HRS9531 injection Placebo — single dose
  Arms: Treatment group E; Treatment group F; Treatment group G; Treatment group H

SUMMARY:
To evaluate the efficacy and dose-response relationship of HRS9531 injection versus placebo in controlling blood glucose after 20 weeks of treatment in subjects with type 2 diabetes who have suboptimal glycaemic control after conventional lifestyle or metformin intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ,18-65 years of age, agreed and signed the informed consent
2. Type 2 diabetes mellitus diagnosed for at least 6 months before the screening visit.
3. Treated with conventional lifestyle intervention and stable treatment with metformin (≥1000 mg/day) at least 8 weeks prior to screening.
4. HbA1c 7.5-10.5% (both inclusive) at screening visit.

Exclusion Criteria:

1. Presence of any clinically significant results in examination at screening visit.
2. Uncontrollable hypertension.
3. A history of type 1 diabetes, specific diabetes, or secondary diabetes.
4. Acute diabetic complications or severe hypoglycemia events within 12 months prior to screening.
5. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening.
6. Any organ-system malignancies developed within 5 years except for cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.
7. Present or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other more serious mental illness.
8. Surgery is planned during the trial.
9. Mentally incapacitated or speech-impaired.
10. Pregnant or lactating woman.
11. In the investigator's judgment, there were circumstances that affected subject safety or otherwise interfered with the evaluation of results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c after 20 weeks of treatment | Week 0 to Week 20

SECONDARY OUTCOMES:
Proportion of subjects reaching HbA1c targets (HbA1c<7.0%) after 20 weeks of treatment | Week 0 to Week 20
Proportion of subjects reaching HbA1c targets (HbA1c<7.0%) after 32 weeks of treatment | Week 0 to Week 32
Change From Baseline in HbA1c after 32 weeks | Week 0 to Week 32
Change from baseline in fasting plasma glucose (FPG), serum insulin and C-peptide after 20 weeks of treatment | Week 0 to Week 20
Change from baseline in fasting plasma glucose (FPG), serum insulin and C-peptide after 32 weeks of treatment | Week 0 to Week 32
Change from baseline body Weight and waist circumference after 20 weeks of treatment | Week 0 to Week 20
Change from baseline in body Weight and waist circumference after 32 weeks of treatment | Week 0 to Week 32
Number of Participants With Anti-HRS9531 Antibody | Week 0 to Week 36
Number of AEs During the Trial | Week 0 to Week 36

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided